CLINICAL TRIAL: NCT02045342
Title: The Effect of a Carbohydrate Drink on Cognitive Function and Exercise Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 104111
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carbohydrate drink (Experimental): Ingest 500ml (1g/kg) prior to metabolic measures.
  Interventions: Other: Carbohydrate drink; Other: Placebo
- Placebo (Placebo Comparator): Ingest 500ml of placebo prior to metabolic measures.
  Interventions: Other: Carbohydrate drink; Other: Placebo

INTERVENTIONS:
Other: Carbohydrate drink — Ingest 500ml (1g/kg) prior to metabolic measures.
Other: Placebo — Ingest 500ml of placebo prior to metabolic measures.

SUMMARY:
This study will investigate the effects of hydrothermally modified starch (SuperStarch) in adults. SuperStarch, originally developed as a drink for children with glycogen storage disease, is a slow digestible carbohydrate, maintaining blood sugar levels over extended periods. Therefore, it could be beneficial to exercise and mental performance, and could possibly have fat loss effects by increasing feelings of fullness. In this study, measures will be taken in 25 men to assess mental function, appetite, and metabolism to determine the processes involved in possible fat loss.

ELIGIBILITY:
Inclusion Criteria:

* healthy, 18 to 35 year old man or woman.

Exclusion Criteria:

* smoker
* pregnancy
* taking part in other research.
* followed a weight loss diet in the previous 6 months.
* history of gastrointestinal, endocrine, cardiovascular disease or diabetes.
* neurological or psychiatric condition that may cause cognitive dysfunction.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Oxygen Consumption | Four 10 minute measures throughout 90 min protocol (1 day).

SECONDARY OUTCOMES:
Appetite ratings | Four appetite ratings throughout 90 min protocol (1 day).
Cognitive function | 2 computerized tests (Stroop Test, Trail Making test) repeated 3 times throughout 90 min protocol (1 day).

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Nutrition Research Laboratory, Western University, London, Ontario, Canada